CLINICAL TRIAL: NCT06641440
Title: Prednisone Plus Levothyroxine Versus Only Levothyroxine to Treat RPL and RIF Women With Thyroisd Autoimmunity Positive to Embryotoxicity Test.
Brief Title: Treatment With Prednisone of Women With RPL or RIF Positive to Antithyroid Antibodies and Embryotoxicity Test
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre for Endocrinology and Reproductive Medicine, Italy (Network)
Responsible Party: Principal Investigator, Fabio Scarpellini, MD, PhD, Centre for Endocrinology and Reproductive Medicine, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CH-06-18
Record Dates: First submitted 2024-10-12; First posted 2024-10-15 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Recurrent Pregnancy Loss, Not Pregnant; Recurrent Implantation Failure
Keywords: antithyroid antibodies; RPL; RIF; embryotoxicity test; predisone treatment; levothyroxine
MeSH Terms: interventions — Prednisone; Thyroxine

STUDY DESIGN:
Intervention Model Description: 25 mg prednisone plus 75 microgram levothyroxine daily 75 micrograms levothyroxine daily
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prednisone plus levothyroxine (Experimental): 25 mg of predisone plus 75 microgram levothyroxine daily for 3 months
  Interventions: Drug: Prednisone
- levothyroxine only (Active Comparator): 75 micrograms of levothyroxine only daily for three months
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Prednisone — patients will be treated for three months in the two groups with the two different protocols for three months both
  Other Names: levothyroxine

SUMMARY:
In Reproductive Medicine there is a unresolved question, whether thyroid autoimmunity may promote infertility, embryo demise and miscarriage. A study was conducted in order to evaluate which treatment is more effective in women with recurrent pregnancy loss (RPL) or recurrent implantation failure (RIF) and positivity to anti-thyroid antibodies to improve their livebirth rate. The patients were treated with prednisone plus levothyroxine in the study group, whereas in the control group the women were treated only with levothyroxine. The patients were treated at least three months before to try again to remain pregnant in case of RPL or to undergo to another embryo transfer with a single blastocyst in case of RIF. The patients during treatment and during the eventual pregnancy will followed up with beta-HCG, anti-thyroid antibodies and TSH levels, as well as ultrasound scan to evaluate the embryo growth and its wellbeing. A statistical analysis will be performed to determine the levels of significance for the parameters evaluated.

DETAILED DESCRIPTION:
This controlled study follows our observational study where we evaluated the frequency of positivity of patients with RPL or RIF to antithyroid antibodies and at the same time their positivity to the embryotoxicity test. In the observational study we documented how a high percentage of these women were positive for antithyroid antibodies, more than 20%, and at the same time these women were also positive to the embryotoxicity test (more than 80% of patients positive for antithyroid antibodies were also positive for the embryotoxicity test). Consequently we decided to conduct a controlled study on the treatment of these patients, all euthyroid, with corticosteroids, predisone, plus levothyroxine comparing them to similar patients treated with levothyroxine only. The study will be conducted in patients with unexplained RPL (3 or more pregnancies lost before the 20th week, without any recognized cause for RPL, such as uterine anomalies, parental chromosomal abnormalities, genetic or acquired thrombophilia) or with unexplained RIF (patients who failed to become pregnant after the transfer of at least 4 good quality blastocysts, without recognized cause for RIF according to the scientific literature). The patients will be randomly assigned, by a computer generated sequency to one of the two arms of the study, the study group where the patients included will be treated with 25 mg of Prednisone plus 75 micrograms of Levothyroxine for at lest three months, and the women included in the control will be treated with 75 micrograms of Levothyroxine for at lest three months, similarly to other group.Afterwards, women will be tested for thyroid antibodies (anti-thyroglobulin and anti-thyroid peroxidase) and for embryotoxicity test. Patients will be able to plan a pregnancy after this in case of RPL or for an embryo transfer with a previously cryopreserved blasocyst.. The sample size calculation for an increase of 100% of the anticipated success rate (livebirth rate as primary end point) in the control group of 30% in bothh type of patients with RPL and RIF showed the needs of 42 patients for arm to have an alfa of <0.05 and a power of 0.8. The primary outcome will be the livebirth rate, and secondary outcome will be pregnancy rate for RIF, abortion rate and negativization rate of the thyroid antibodies and embryotoxicity test.

ELIGIBILITY:
Inclusion Criteria:

* euthyroid women
* with RPL
* with RIF, positivity to anti-thyroid antibodies (anti thyreoglobulin and/or anti thyroid peroxidase),

Exclusion Criteria:

* No autoimmune diseases (SLE, RA),
* no diabetes,
* no hearth diseases,
* no egg donation cases,

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — only women
Enrollment: 42 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
livebirth rate | all the study time 5 yeard time frame
  number of babyis born divided the number become pregnant

SECONDARY OUTCOMES:
pregnancy rate | all the study time 5 yeard time frame
  the number of women become pregnant divided for all women included in the study
abortion rate | all the study time 5 yeard time frame
  the number of abortion divided the number of pregnancy
the negativization rate of antithyroid antibodies | all the study time 5 yeard time frame
  number of patients positive for thyroid antibodies who become negative percent

CONTACTS AND LOCATIONS:
Overall Officials: Daniela A Marconi, MD, Study Chair — Centre for Endocrinology and Reproductive Medicine, Italy
Locations (2):
- Italy (2):
  - CERM-Hungaria IVF Center, Rome, RM
  - Cerm-Hungaria, Rome

IPD SHARING:
Plan to Share IPD: No